CLINICAL TRIAL: NCT04551508
Title: Delirium Screening 3 Methods Study (DELIS-3). Agreement Between CAM-ICU, CAM-ICU-7 and ICDSC in a Danish Population of ICU Patients and Nurses' Perception of the Clinical Relevance of Delirium Screening
Brief Title: Delirium Screening 3 Methods Study
Acronym: DELIS-3
Status: Completed | Type: Observational
Sponsor: Hospitalsenheden Vest (Other)
Responsible Party: Principal Investigator, Anne Højager Nielsen, Principal Investigator, MCN, PH.D., Hospitalsenheden Vest
Other Study IDs: 31-1521-440 (STPS)
Record Dates: First submitted 2020-09-09; First posted 2020-09-16 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Delirium; Critical Illness
MeSH Terms: conditions — Delirium; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Observational study comparing three different methods of delirium detection in critically ill patients.

DETAILED DESCRIPTION:
The DELIS-3 study aims to compare three different approaches to detection of ICU (intensive care unit) delirium in critically ill patients. The CAM-ICU (Confusion Assessment Method for the ICU) and the ICDSC (Intensive Care Delirium Screening Checklist) have both been developed in the early 1990. The CAM-ICU is either positive or negative, whereas the ICDSC is a score between 0-8. A score above 3 is delirium positive. Neither scale has been validated as severity scales. The novel CAM-ICU-7 is developed from the original CAM-ICU and has been validated as a severity scale.

Detection of delirium in critically ill patients is highly necessary as delirium can be very painful to the patient. Moreover, certain subtypes of delirium is associated with increased mortality and poorer cognitive outcome when patients are followed up on long term.

Therefore, delirium screening of all patients is standard care in most intensive care units.

However, there is also a need to assess severity of delirium. The recently published CAM-ICU-7 has now been translated to Danish and this study will explore its performance compared to the CAM-ICU and the ICDSC.

In 17 Danish ICU's 10 nurses will be trained in using all three instruments. Each nurse will subsequently screen 10 patients each with all three instruments as part of their normal practice. The sequence of the instruments will be randomized to avoid that one instrument is favored by always being used first, second or last.

For each patient the following data will be collected: sex, age, reason for hospitalization (medical, neurological, surgical/ acute, planned), ventilator treatment, ability to verbalize, RASS score (sedation and agitation score) severity of disease (SMS score) and time of admission.

After all screenings has been collected, nurses will fill in a questionnaire on their perceptions of each scales' ability to reliably detect delirium, userfriendliness and how time consuming each scale were to use.

ELIGIBILITY:
Inclusion Criteria:

* All patients admitted to critical care units.

Exclusion Criteria:

* Patients with RASS score of -3, -4, -5

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients admitted to critical care units may be included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 1126 (Actual)
Dates: Start 2020-09-09 (Actual); Primary Completion 2021-11-01 (Actual); Study Completion 2021-11-01 (Actual)

PRIMARY OUTCOMES:
Confusion Assessment Method of the Intensive Care Unit (CAM-ICU) | Day 1
  Clinical test for detecting delirium bedside, can be used by non-psychiatrists. CAM-ICU can be either positive (indicating delirium) or negative.
Confusion assessment method of the intensive care unit 7 (CAM-ICU -7) | Day 1
  Clinical test for detecting delirium bedside, can be used by non-psychiatrists. CAM-ICU-7 can yield a score of 0-7 points, higher values indicative of worse delirium.
intensive care delirium screening checklist (ICDSC) | Day 1
  Clinical test for detecting delirium bedside, can be used by non-psychiatrists. ICDSC can yield a score of 0-8 points, higher values indicative of worse delirium.

CONTACTS AND LOCATIONS:
Overall Officials: Helle Svenningsen, ph.d., Principal Investigator — VIA University College, Aarhus, Denmark
Locations (14):
- Denmark (14):
  - Regionshospitalet Herning, Herning, Central Jutland
  - Regionshospitalet Holstebro, Holstebro, Central Jutland
  - Odense Universitetshospital, Odense, C
  - Aalborg Universitetshospital, Aalborg
  - Aarhus Universitetshospital, Aarhus
  - Rigshospitalet, Copenhagen Ø
  - Sydvestjysk sygehus, Esbjerg
  - Nordsjællands Hospital, Hillerød
  - Holbæk Sygehus, Holbæk
  - Regionshospitalet Horsens, Horsens
  - Sjællands Universitetshospital, Køge
  - Regionshospitalet Randers, Randers
  - Vejle Sygehus, Vejle
  - Regionshospitalet Viborg, Viborg

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Khan BA, Perkins AJ, Gao S, Hui SL, Campbell NL, Farber MO, Chlan LL, Boustani MA. The Confusion Assessment Method for the ICU-7 Delirium Severity Scale: A Novel Delirium Severity Instrument for Use in the ICU. Crit Care Med. 2017 May;45(5):851-857. doi: 10.1097/CCM.0000000000002368. PMID 28263192
- [Background] Bergeron N, Dubois MJ, Dumont M, Dial S, Skrobik Y. Intensive Care Delirium Screening Checklist: evaluation of a new screening tool. Intensive Care Med. 2001 May;27(5):859-64. doi: 10.1007/s001340100909. PMID 11430542
- [Background] Ely EW, Margolin R, Francis J, May L, Truman B, Dittus R, Speroff T, Gautam S, Bernard GR, Inouye SK. Evaluation of delirium in critically ill patients: validation of the Confusion Assessment Method for the Intensive Care Unit (CAM-ICU). Crit Care Med. 2001 Jul;29(7):1370-9. doi: 10.1097/00003246-200107000-00012. PMID 11445689
- [Background] Almgren M, Lundmark M, Samuelson K. The Richmond Agitation-Sedation Scale: translation and reliability testing in a Swedish intensive care unit. Acta Anaesthesiol Scand. 2010 Jul;54(6):729-35. doi: 10.1111/j.1399-6576.2009.02173.x. Epub 2009 Dec 5. PMID 20002362
- [Background] Granholm A, Perner A, Krag M, Marker S, Hjortrup PB, Haase N, Holst LB, Collet MO, Jensen AKG, Moller MH. External validation of the Simplified Mortality Score for the Intensive Care Unit (SMS-ICU). Acta Anaesthesiol Scand. 2019 Oct;63(9):1216-1224. doi: 10.1111/aas.13422. Epub 2019 Jul 4. PMID 31273763